CLINICAL TRIAL: NCT05205577
Title: Trial of Auricular Vagus Nerve Stimulation in Painful Covid Long
Acronym: COLOSAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Schwa medico (device lending) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: APHP211364; IDRCB 2021-A00874-37 (Other: ANSM)
Record Dates: First submitted 2022-01-24; First posted 2022-01-25 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: long covid; pain; Neuromodulation
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tens Eco Plus — 30min/day of stimulation at 25Hz frequency, 100 microsc pulse with intensity escalation up to 25 mA max

SUMMARY:
Patients infected with Covid 19 suffer from frequent pain (headache, migraines, joint pain, muscle pain) in the acute phase which may persist after a stay in intensive care or in an intensive care unit, in the event of post-traumatic stress syndrome, pre-existing comorbidities.

The pain mechanisms observed during the covid epidemic are nociceptive / inflammatory pain, neuropathic pain, and nociplastic pain.

Auricular transcutaneous vagus nerve stimulation (tVNS) is a promising therapeutic strategy that may reduce inflammation and pain level.

Colosat is a prospective non-randomized pilot feasibility study. Colosat is a 8 weeks non randomized trial investigating the painful Covid long.

tVNS will be performed using a transcutaneous lectrical nerve stimulation (TENS) device connected to an auricular electrode stimulating the cutaneous area of the left ear innervated by the auricular ascendant branch of the vagus nerve.

DETAILED DESCRIPTION:
Covid-19 is a disease that presents in several clinical forms (severity and duration). From the end of the first epidemic wave in May 2020, the persistence of symptoms several weeks or months after the first manifestations were described in more than 20% of patients after 5 weeks and more and in more than 10% of patients after 3 months.

In the acute phase, the pains are frequent: headaches / migraines about 13%, joint pain 15%, muscle pain 36%.

In the longer term, patients infected with the coronavirus whose condition necessitated a stay in intensive care have an increased risk of having sequelae (nociceptive or neuropathic) pain. A study carried out 2 years after a stay in an intensive care unit on 164 patients showed that 56% of them suffered from chronic pain. A retrospective study of 80 patients who were hospitalized in the intensive care unit for acute respiratory distress syndrome showed that 38% of them suffered from chronic pain. A meta-analysis of 9 studies and including 1419 patients shows that the incidence or prevalence of pain 3 months after discharge from the intensive care unit ranges from 28 to 77%.

Many viral infections induce neuropathic pain such as Guillain Barré syndrome with an estimated prevalence of 0.5 to 1% and more complex pain syndromes, some of which may suggest nociplastic pain (pain without lesion as in fibromyalgia). There is also a risk of painful chronicization, in particular in the event of post-traumatic stress and / or anxiety-depressive disorders and pre-existing comorbidities (anxiety-depression) There are several pain mechanisms observed during the covid epidemic: nociceptive / inflammatory pain, neuropathic pain, nociplastic pain (without injury).

Pain management is medication with the prescription of analgesics according to the classification of the International Association for the Study of Pain according to the pain-generating mechanism as well as non-drug therapeutic approaches.

Transcutaneous electrical neurostimulation is an analgesic method widely used in Pain Assessment and Treatment Centers in addition to drug analgesics.

The vagus nerve (belonging to the parasympathetic system) is the cranial nerve whose territory is the most extensive having several functions (slowing the heart rate, promoting digestion, improving sleep, etc.). It is a mixed nerve comprising 80% afferent fibers and 20% efferent fibers. It has anti-inflammatory properties both via its afferent fibers capable of activating the corticotropic axis in response to immune stress and, more recently, via its efferent fibers. The release of acetylcholine at the end of its efferent fibers is able to inhibit the release of pro-inflammatory cytokines from splenic macrophages.

This anti-TNF property of the vagus nerve has been used in the treatment of chronic inflammatory bowel diseases but also in rheumatoid arthritis. Any abnormality of the sympathovagal balance can have a pro-inflammatory effect. The reestablishment of this sympathovagal balance is therefore likely to counterbalance a pro-inflammatory process.

In addition, stress also plays a role as it causes vagal inhibition and activation of the sympathetic system thereby promoting the pro-inflammatory reaction. Depending on the environment and the circumstances, stimulation of the vagus nerve can help the body to find the right balance between the sympathetic and parasympathetic systems and therefore a good sympathovagal balance.

Stimulation of the vagus nerve by implantable device, authorized for refractory depression or epilepsy. It has also been considered for several years to treat pain. For pain, a study of 14 patients with fibromyalgia showed a decrease in pain sensitivity corroborated by QST (Quantitative Sensory Testing) before stimulation and at 4, 6, 9 and 12 months after. The use of an implantable device is invasive and is not used in routine practice (surgery).

Functional MRI studies have shown that minimally invasive and inexpensive transcutaneous atrial electrical stimulation (tVNS) (of the left cymba concha) activates the central vagal centers.

However, this stimulation technique (unlike TENS) has been little evaluated for treating pain (3 randomized controlled clinical trials). For induced experimental pain (mechanical pain, pressure pain, thermal pain), atrial tVNS at 25 Hz increased the threshold for mechanical pain and pressure and reduced sensitivity to mechanical pain in 48 healthy subjects (trial controlled cross over). In chronic migraine, a randomized controlled study including 46 patients showed a reduction in the frequency of headaches for 13 to 29% of them depending on the stimulation groups (25Hz versus 1Hz). Another open multicenter study on 50 patients showed a reduction in pain in 64.6% of patients.

tVNS can be performed effectively using a transcutaneous electrical nerve stimulation (TENS) machine. In this case, the TENS machine is coupled to an atrial electrode designed to apply anatomically to contact with the cymba concha in the left ear to avoid parasympathetic cardiovascular effects when stimulated in the right ear.

We want to set up a pilot clinical study to assess the value of this non-drug therapeutic strategy in the overall management of pain from long-term COVIDs. The objective is to have a 1st evaluation of the efficacy, tolerance and feasibility of transcutaneous atrial vagus nerve stimulation (tVNS) in the various pain mechanisms (nociceptive, neuropathic and nociplastic) observed during the Covid-19. Depending on the results, a randomized controlled trial may then be set up. ?

Colosat is a 8 weeks non randomized trial investigating the painful Covid long. tVNS will be performed using a transcutaneous lectrical nerve stimulation (TENS) device connected to an auricular electrode stimulating the cutaneous area of the left ear innervated by the auricular ascendant branch of the vagus nerve.

ELIGIBILITY:
Inclusion Criteria:

Subjects aged 18 to 80 with prolonged post-Covid-19 pain defined by 3 criteria according to the Haute Autorité de Santé :

* Symptomatic initial episode of Covid-19 is confirmed by at least one criterion among: PCR SARS-CoV-2 +, antigenic test SARS-CoV-2 +, Serology SARS-CoV-2 +, prolonged anosmia / ageusia of sudden onset , chest scanner
* Presence of at least one of the initial symptoms, beyond 4 weeks following the onset of the acute phase of the disease
* Initial and prolonged symptoms not explained by another diagnosis with no known link to Covid-19

  * With intact and uninjured skin at the level of the cymba concha of the left ear
  * Signature of informed consent
  * Pain of intensity> or equal to 40 mm / 100mmm on the Visual Analogue Scale (VAS) over the last 7 days before inclusion, analgesic treatment stable for at least 2 weeks
  * Must be able to comply with protocol requirements
  * Beneficiary of a social security scheme or entitled

Exclusion Criteria:

* Having a hearing aid device with a left cochlear implant
* Having a major hearing loss
* Having an unsuitable ear canal
* Use of other electrically active medical devices (TENS for chronic pain, pacemaker)
* Taking treatment with strong opioids, corticosteroids or nonsteroidal anti-inflammatory drugs systemically (oral, subcutaneous, intravenous, intramuscular, transdermal).
* With cognitive disorders that do not allow answering questionnaires and /or setting up the device
* Known history of cardiac arrhythmias, atrioventricular block> 1st degree, conduction disorders
* Symptomatic orthostatic hypotension or history of recurrent vagal syncope
* History of vagotomy
* severe asthma
* Pregnant, breastfeeding or having a desire to become pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain | 2 months
  Difference D0-M2 of self-reported pain post Covid-19 (COVID Long) measured in a 100 mm on a Visual Analog Scale (VAS).
  The patient assesses the pain of the last eight days before the visit.

SECONDARY OUTCOMES:
Analgesics | 2 months
  consumption of analgesics during visits on D0 and M2 (modification of doses)
PGIC | 2 months
  Patient global impression of change at M2
Quality of life | 1 and 2 months
  improvement of the quality of life between Do and M2
Side effects | 1 and 2 months
  report of side effects during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Mauboussin Carlos, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Centre d'Evaluation et de Traitement de la Douleur, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided